CLINICAL TRIAL: NCT01270165
Title: Antiviral Efficacy of Continuing Lamivudine Plus Adefovir or Switching to Telbivudine Plus Adefovir in HBeAg-positive Lamivudine-refractory Chronic Hepatitis B Patients Who Have Suboptimal Response to Lamivudine Plus Adefovir for at Least 12 Months
Brief Title: Lamivudine Plus Adefovir Versus Telbivudine Plus Adefovir in Lamivudine Resistant Chronic Hepatitis B
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2010-0168
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Hepatitis B
Keywords: lamivudine; telbivudine; adefovir; lamivudine resistance
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: telbivudine — 600mg, oral daily over 12 months

SUMMARY:
No study has reported on the comparative effect of continuing lamivudine plus adefovir versus switching to telbivudine plus adefovir in HBeAg-positive lamivudine-refractory chronic hepatitis B patients who have suboptimal response to lamivudine plus adefovir. The goal of this study is to compare the efficacy of continuing lamivudine plus adefovir versus switching to telbivudine plus adefovir directly in patients with lamivudine-refractory chronic hepatitis B patients who have suboptimal response to lamivudine plus adefovir for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg positive
* lamivudine and adefovir at least 12 months over 6 months lamivudine treatment for YMDD positive patients
* HBV DNA over 300 copies/ml

Exclusion Criteria:

* decompensated cirrhosis
* renal failure
* prior interferon usage
* evidence of HCC or prior organ transplantation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Virologic response | 1 year

SECONDARY OUTCOMES:
Safety, virologic breakthrough and biochemical response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, MD, PhD, Principal Investigator — Department of Internal Medicine, Yonsei University College of Medicine
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park H, Park JY, Kim SU, Kim DY, Han KH, Chon CY, Ahn SH. Efficacy of switching to telbivudine plus adefovir in suboptimal responders to lamivudine plus adefovir. World J Gastroenterol. 2013;19(43):7671-9. doi: 10.3748/wjg.v19.i43.7671. PMID 24431895